CLINICAL TRIAL: NCT05567341
Title: Remote Ischemic Preconditioning in Vestibular Schwannoma Surgery and Its Neuroprotective Effect on the Cochlear and Facial Nerve Function
Brief Title: Remote Ischemic Preconditioning in Vestibular Schwannoma Surgery
Acronym: RIC-VS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 489-0-0
Record Dates: First submitted 2022-09-26; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Vestibular Schwannoma
Keywords: remote ischemic preconditioning; cochlear nerve; facial nerve; hearing; vestibular schwannoma surgery
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Intervention Model Description: group 1: intervention, remote ischemic preconditioning for 4x5 minutes at the beginning of the surgery group 2: sham-control (4x5 min without compression of the extremity)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: only the study nurse who performs the intervention is aware of the study arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC (Experimental): On the right upper extremity a blood pressure cuff is inflated to 200mmHg for 4x5min at the beginning of the surgery
  Interventions: Procedure: Remote ischemic preconditioning
- Control (Sham Comparator): On the right upper extremity a blood pressure cuff is inflated to 0mmHg for 4x5min at the beginning of the surgery
  Interventions: Procedure: Sham-control

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — A blood pressure cuff is inflated to 200 mmHg for 4x5 min (5 min rest between cycles) at the right upper extremity when the vestibular schwannoma surgery is started
  Arms: RIC
Procedure: Sham-control — A blood pressure cuff is inflated to 0 mmHg for 4x5 min (5 min rest between cycles) at the right upper extremity when the vestibular schwannoma surgery is started
  Arms: Control

SUMMARY:
Vestibular schwannomas are primarily benign (WHO grade I) tumors originating from the Schwann cells of the vestibular nerve and are among the most common tumors of the skull base. Common treatment options are surgical tumor resection or targeted radiation therapy. The special challenge of surgical treatment is the functional preservation of the cranial nerves, especially the cochlear and facial nerves. Perioperative ischemia of the cochlea and cochlear nerve is postulated as the underlying mechanism of postoperative hearing loss. Ischemic preconditioning is a non-invasive procedure that triggers the release of vasoactive cytokines and mediators by repeated short-term induction of limb ischemia. Improved perfusion of critically perfused end organs as well as a reduction of cerebral infarct volumes has already been shown in other pathologies. In the planned study, possible neuroprotective effects of remote ischemic preconditioning on postoperative hearing as well as facial nerve function in patients with vestibular schwannomas will be examined.

DETAILED DESCRIPTION:
Purpose: Does remote ischemic preconditioning improve hearing and/or facial nerve palsy after resection of vestibular schwannomas?

Study Design: Prospective, randomized, double-blind, single-center.

Case number: The study should include 120 patients (60 treatment arm, 60 control arm). Case number calculation (mean effect sizes, chi-square test, alpha error = 0.05, beta error = 20%) results in a necessary total patient number of 100 with 50 patients per group. Including the expected dropout rate (approx. 20%), the required total number of study participants is set at 120 patients. With approximately 55 patients/year in whom anatomic preservation of the cochlear nerve is possible intraoperatively, the total study duration is estimated to be approximately 2-2.5 years.

Study procedure: Day 1

* Preoperative pure tone audiometry including speech discrimination and preoperative AEP measurement
* preoperative assessment of facial nerve function according to House and Brackmann and photo documentation
* Preoperative blood sample (Hg, WBC, platelet count, creatinine, sodium, potassium, CRP, PCT, IL-6, INR, Quick, aPTT, d-dimer)
* Evaluation of inclusion and exclusion criteria, informed consent

Day 2

* Randomization
* At skin incision RIC procedure or sham control.

  * RIC arm: 5 minutes inflation of a blood pressure cuff to 200mmHg on the right arm, then 5 minutes rest, the procedure will be performed 4 times in total.
  * Control arm: 5 minutes inflation of a blood pressure cuff to 0mmHg on the right arm, then 5 minutes rest, the procedure will be performed 4 times in total.
* Performance of tumor resection under electrophysiological monitoring.
* blood sample (Hg, WBC, platelet count, creatinine, sodium, potassium, CRP, PCT, IL-6, INR, Quick, aPTT, d-dimer)

Day 3

* blood sample (Hg, WBC, platelet count, creatinine, sodium, potassium, CRP, PCT, IL-6, INR, Quick, aPTT, d-dimer)
* Clinical assessment of facial nerve function
* Evaluation of complications

Before discharge

* Clinical assessment of facial nerve function and photo documentation
* Evaluation of complications occurring in the course of the procedure
* Postoperative AEP measurement and pure tone audiometry incl. speech discrimination

Outpatient follow-up after 3 months

* Evaluation of postoperative pure tone audiometry incl. speech discrimination
* Clinical assessment of facial nerve function and photo documentation

Objective:

Primary outcome: patients undergoing RIC will show better hearing 3 months postoperatively than the sham control group.

Secondary outcome hypothesis: patients undergoing RIC will show better postoperative facial nerve function than the sham control group before discharge and 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* total or gross-total resection of a vestibular schwannoma is planned
* Functional hearing is still present on the affected side preoperatively (AEP evocable and Gardner-Robertson grade I, II, or III).
* Preoperatively, facial function is unimpaired or mildly impaired (House and Brackmann grade I or II).

Exclusion Criteria:

* Symptomatic peripheral artery disease.
* Active or previous thrombosis in the extremity where the RIC procedure is to be performed.
* Neurofibromatosis type 2
* Only planned decompression of the internal auditory canal without relevant tumor resection
* Pregnant or breastfeeding females
* Previous radiotherapy of the vestibular schwannoma that will be resected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
postoperative hearing | 3 months (± 6 weeks) after surgery
  hearing on pure tone audiometry according to AAO-HNS/Gardner-Robertson

SECONDARY OUTCOMES:
postoperative facial nerve function | up to 8 days after surgery
  facial nerve function according to House and Brackmann
postoperative facial nerve function | 3 months (± 6 weeks) after surgery
  facial nerve function according to House and Brackmann

OTHER OUTCOMES:
postoperative hearing | up to 8 days after surgery
  hearing on pure tone audiometry according to AAO-HNS/Gardner-Robertson
laboratory findings | within 4 hours after surgery
  White blood count
laboratory findings | within 4 hours after surgery
  C-reactive protein
laboratory findings | within 4 hours after surgery
  Procalcitonin
laboratory findings | within 4 hours after surgery
  Interleukin 6
laboratory findings | within 4 hours after surgery
  D-Dimer
laboratory findings | within 4 hours after surgery
  platelet count
laboratory findings | within 4 hours after surgery
  International normalized ratio (INR)
laboratory findings | within 4 hours after surgery
  activated partial thromboplastin time (aPTT)
laboratory findings | postoperatively, 1 day after surgery
  White blood count
laboratory findings | postoperatively, 1 day after surgery
  C-reactive protein
laboratory findings | postoperatively, 1 day after surgery
  Procalcitonin
laboratory findings | postoperatively, 1 day after surgery
  Interleukin 6
laboratory findings | postoperatively, 1 day after surgery
  D-Dimer
laboratory findings | postoperatively, 1 day after surgery
  platelet count
laboratory findings | postoperatively, 1 day after surgery
  International normalized ratio (INR)
laboratory findings | postoperatively, 1 day after surgery
  activated partial thromboplastin time (aPTT)
postoperative AEP | up to 8 days after surgery
  Auditory evoked potentials after surgery
postoperative vertigo | up to 8 days after surgery
  Vertigo according to dizziness handicap inventory (=DHI, score 0-100, higher scores are associated with a higher burden of dizziness)
postoperative vertigo | 3 months (± 6 weeks) after surgery
  Vertigo according to dizziness handicap inventory (=DHI, score 0-100, higher scores are associated with a higher burden of dizziness)
extent of schwannoma resection | 3 months (± 6 weeks) after surgery
  extent of schwannoma resection on the postoperative MRI

CONTACTS AND LOCATIONS:
Overall Officials: Contantin Roder, Prof., MD, Principal Investigator — Department of Neurosurgery Tuebingen; Helene V Hurth, MD, Principal Investigator — Department of Neurosurgery Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
IPD may be shared on request after completion of the study and as soon as data will be published.